CLINICAL TRIAL: NCT04686721
Title: A Retrospective and Prospective Observational, Multicentric, Case-control Clinical Study for the Evaluation of Tracheal Stenosis Among Patients With COVID-19 and Prolonged Intubation or Tracheostomy.
Brief Title: Observational Study for the Evaluation of Tracheal Stenosis in COVID-19 Patients
Acronym: TS1
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istituto Clinico Humanitas (Other)
Responsible Party: Sponsor
Other Study IDs: TS1
Record Dates: First submitted 2020-12-21; First posted 2020-12-29 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Tracheal Stenosis
Keywords: Tracheal Stenosis; COVID-19; Prolonged intubation; Tracheostomy; SARS-CoV-2
MeSH Terms: conditions — Tracheal Stenosis; COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 8 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients at risk of developing tracheal stenosis after prolonged intubation or tracheostomy: Patients older than 18 years of age who underwent either prolonged intubation or tracheostomy will be enrolled. A minimum of 2 months follow-up from hospital discharge is required. Patients tested negative for SARS-CoV-2 will be used as a control group
  Interventions: Diagnostic Test: Chest CT scan + baseline spirometry

INTERVENTIONS:
Diagnostic Test: Chest CT scan + baseline spirometry — Patients will perform an initial evaluation at 2 months from hospital discharge using a chest CT scan without contrast-enhancing along with a pulmonary function test using spirometry. Based on results and according to current guidelines, further follow-up or intervention will be administered.

SUMMARY:
Define the actual incidence of tracheal stenosis in patients who underwent either prolonged intubation or tracheostomy and to compare incidence, clinical course and outcome between COVID-19 and non-COVID-19 patients.

DETAILED DESCRIPTION:
The TS1 is a national observational, multicentric, case-control clinical aiming at defining the actual incidence of tracheal stenosis in patients with COVID-19 that underwent prolonged intubation or tracheal stenosis.

Information regarding anamnestic data, demographics, smoking or alcohol habits, comorbidity, previous history of prolonged ventilation or tracheostomy, and data about intensive care unit stay and treatment will be collected before discharging patients from hospital.

All patients enrolled will perform an initial evaluation with a chest CT scan without contrast-enhancing at 2 months from hospital discharge along with pulmonary function test. If tracheal stenosis is detected, treatment according to currently available guidelines will be performed.

Patients with no signs of clinical, functional and radiological evidence of tracheal stenosis will perform a 3 and 6 months clinical follow-up from initial evaluation.

A chest CT scan with pulmonary function test will be administered if symptoms of tracheal stenosis arise during clinical follow-up. If necessary, treatment according to currently available guidelines will be performed.

Patients will be followed-up for 8 months after hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* prolonged intubation, defined as the permanence of naso or oro- tracheal tube for more than 7 days
* tracheostomy, whether surgical or percutaneous
* minimum of 2 months follow-up from hospital discharge
* Positivity to SARS-CoV-2 infection confirmed using PCR on either nasal swab or bronchoalveolar lavage will be not an inclusion criterion; patients tested negative will be used as a control group

Exclusion Criteria:

* Pediatric patients (< 18 years of age)
* Patients without a minimum of 2 months follow-up from hospital discharge

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is addressed to an adult population (> 18 years of age) and will enroll subjects who underwent prolonged intubation or tracheostomy. Patient data collection will be divided in two cohorts:
  * a retrospective cohort admitted to intensive care unit (ICU) from 21/02/2020 to 30/11/2020
  * a prospective cohort will include patients admitted to ICU from 01/12/2020
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-12-20 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of tracheal stenosis following either prolonged intubation or tracheostomy in COVID-19 patients | 8 months
  Observe how many subject in the population at risk will develop tracheal stenosis during follow-up
Clinical presentation of tracheal stenosis | 8 months
  Describe symptoms most commonly associated with tracheal stenosis
Clinical course of tracheal stenosis | 8 months
  Analyse the clinical evolution of tracheal stenosis during follow-up
Outcome of tracheal stenosis | 8 months
  Collect data on morbidity and mortality of tracheal stenosis

SECONDARY OUTCOMES:
Identification of demographic factor with a predictive and prognostic value for tracheal stenosis | 8 months
  Patient's characteristic (e.g. sex, age, weight and height) will be collected during follow-up to search for any statistically significant association with risk of developing tracheal stenosis or disease-free survival
Identification of clinical factor with a predictive and prognostic value for tracheal stenosis | 8 months
  Information regarding hospitalisation (e.g. personal history of diabetes, chronic obstructive pulmonary disease, previous prolonged intubation or tracheostomy) will be collected during follow-up to search for any statistically significant association with risk of developing tracheal stenosis or disease-free survival
Identification of radiological factor with a predictive and prognostic value for tracheal stenosis | 8 months
  Data collected from CT scan performed during follow-up (e.g. distance of stenosis from vocal chords, length and diameter) will be collected during follow-up to search for any statistically significant association with risk of developing tracheal stenosis or disease-free survival
Identification of instrumental factor with a predictive and prognostic value for tracheal stenosis | 8 months
  Results obtained from pulmonary function test (e.g. forced expiratory volume at one second, forced vital capacity and peak expiratory flow rate) will be collected during follow-up to search for any statistically significant association with risk of developing tracheal stenosis or disease-free survival
Compare COVID-19 and non-COVID-19 patients at risk of developing tracheal stenosis | 8 months
  A control-group of patient who underwent either prolonged intubation or tracheostomy without diagnosis of COVID-19 will be used as comparison to search for any difference in primary and secondary outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Humanitas Research Hospital, Rozzano, Italy